CLINICAL TRIAL: NCT03971734
Title: Determining the Dose of Regadenoson Most Likely to Transiently Alter the Integrity of the Blood-Brain Barrier in Patients With High Grade Gliomas
Brief Title: Determining Dose of Regadenoson Most Likely to Transiently Alter the Integrity of the Blood-Brain Barrier in Patients With High Grade Gliomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated [NCI decided to terminate ABTC Consortium due to NCI moving in different direction for Brain Cancer]
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABTC 1804; UM1CA137443 (NIH)
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: High Grade Glioma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Glioblastoma
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Glioblastoma | interventions — regadenoson

STUDY DESIGN:
Intervention Model Description: Seven dose levels of Regadenoson will be studied in part 1, minimum 3 patients per dose level.
  Part 2 will include 5 patients at each level that achieved thresh hold in part 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Arm 1 regadenoson 0.05mg (Experimental): Approximately 10 minutes prior to undergoing the research MRI, patients will be administered a single dose of regadenoson at their assigned dose level, under the supervision of a cardiologist.
  The research MRI scan will be performed immediately following administration of regadenoson and appropriate monitoring of vital signs and 12-lead electrocardiography on a similar machine as the pre-enrollment eligibility MRI scan, using the same administered dose of gadolinium and acquisition parameters.
  The research MRI will consist of DCE perfusion MRI for estimation of Ktrans and will be performed with co-administration of standard doses of gadolinium following regadenoson dose.
  Regadenoson 0.05mg
  Interventions: Drug: Regadenoson 0.05mg
- Arm 2 regadenoson 0.1mg (Experimental): Approximately 10 minutes prior to undergoing the research MRI, patients will be administered a single dose of regadenoson at their assigned dose level, under the supervision of a cardiologist.
  The research MRI scan will be performed immediately following administration of regadenoson and appropriate monitoring of vital signs and 12-lead electrocardiography on a similar machine as the pre-enrollment eligibility MRI scan, using the same administered dose of gadolinium and acquisition parameters.
  The research MRI will consist of DCE perfusion MRI for estimation of Ktrans and will be performed with co-administration of standard doses of gadolinium following regadenoson dose.
  Interventions: Drug: Regadensoson 0.1mg
- Arm 3 regadenoson 0.2mg (Experimental): Approximately 10 minutes prior to undergoing the research MRI, patients will be administered a single dose of regadenoson at their assigned dose level, under the supervision of a cardiologist.
  The research MRI scan will be performed immediately following administration of regadenoson and appropriate monitoring of vital signs and 12-lead electrocardiography on a similar machine as the pre-enrollment eligibility MRI scan, using the same administered dose of gadolinium and acquisition parameters.
  The research MRI will consist of DCE perfusion MRI for estimation of Ktrans and will be performed with co-administration of standard doses of gadolinium following regadenoson dose.
  Interventions: Drug: Regadensoson 0.2mg
- Arm 4 regadenoson 0.4mg (Experimental): Approximately 10 minutes prior to undergoing the research MRI, patients will be administered a single dose of regadenoson at their assigned dose level, under the supervision of a cardiologist.
  The research MRI scan will be performed immediately following administration of regadenoson and appropriate monitoring of vital signs and 12-lead electrocardiography on a similar machine as the pre-enrollment eligibility MRI scan, using the same administered dose of gadolinium and acquisition parameters.
  The research MRI will consist of DCE perfusion MRI for estimation of Ktrans and will be performed with co-administration of standard doses of gadolinium following regadenoson dose.
  Interventions: Drug: Regadensoson 0.4mg
- Arm 5 regadenoson 0.7mg (Experimental): Approximately 10 minutes prior to undergoing the research MRI, patients will be administered a single dose of regadenoson at their assigned dose level, under the supervision of a cardiologist.
  The research MRI scan will be performed immediately following administration of regadenoson and appropriate monitoring of vital signs and 12-lead electrocardiography on a similar machine as the pre-enrollment eligibility MRI scan, using the same administered dose of gadolinium and acquisition parameters.
  The research MRI will consist of DCE perfusion MRI for estimation of Ktrans and will be performed with co-administration of standard doses of gadolinium following regadenoson dose.
  Interventions: Drug: Regadensoson 0.7mg
- Arm 6 regadenoson 1.0mg (Experimental): Approximately 10 minutes prior to undergoing the research MRI, patients will be administered a single dose of regadenoson at their assigned dose level, under the supervision of a cardiologist.
  The research MRI scan will be performed immediately following administration of regadenoson and appropriate monitoring of vital signs and 12-lead electrocardiography on a similar machine as the pre-enrollment eligibility MRI scan, using the same administered dose of gadolinium and acquisition parameters.
  The research MRI will consist of DCE perfusion MRI for estimation of Ktrans and will be performed with co-administration of standard doses of gadolinium following regadenoson dose.
  Interventions: Drug: Regadensoson 1.0mg
- Arm 7 regadenoson 1.4mg (Experimental): Approximately 10 minutes prior to undergoing the research MRI, patients will be administered a single dose of regadenoson at their assigned dose level, under the supervision of a cardiologist.
  The research MRI scan will be performed immediately following administration of regadenoson and appropriate monitoring of vital signs and 12-lead electrocardiography on a similar machine as the pre-enrollment eligibility MRI scan, using the same administered dose of gadolinium and acquisition parameters.
  The research MRI will consist of DCE perfusion MRI for estimation of Ktrans and will be performed with co-administration of standard doses of gadolinium following regadenoson dose.
  Interventions: Drug: Regadensoson 1.4mg

INTERVENTIONS:
Drug: Regadenoson 0.05mg — Regadensoson 0.05mg administered prior to MRI
  Arms: Arm 1 regadenoson 0.05mg
Drug: Regadensoson 0.1mg — Regadensoson 0.1mg administered prior to MRI
  Arms: Arm 2 regadenoson 0.1mg
Drug: Regadensoson 0.2mg — Regadensoson 0.2mg administered prior to MRI
  Arms: Arm 3 regadenoson 0.2mg
Drug: Regadensoson 0.4mg — Regadensoson 0.4mg administered prior to MRI
  Arms: Arm 4 regadenoson 0.4mg
Drug: Regadensoson 0.7mg — Regadensoson 0.7mg administered prior to MRI
  Arms: Arm 5 regadenoson 0.7mg
Drug: Regadensoson 1.0mg — Regadensoson 1.0mg administered prior to MRI
  Arms: Arm 6 regadenoson 1.0mg
Drug: Regadensoson 1.4mg — Regadensoson 1.4mg administered prior to MRI
  Arms: Arm 7 regadenoson 1.4mg

SUMMARY:
enroll patients with histologically confirmed high-grade gliomas to evaluate the ability of regadenoson to transiently disrupt a relatively intact blood-brain barrier (BBB). determine the best dose of regadenoson to disrupt the BBB and allow for enhanced penetration of gadolinium during MRI.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine if there is a dose of regadenoson, in the range shown to be safe for clinical administration, that can increase gadolinium Ktrans by more than 10 times the values reported in the literature within normal-appearing brain parenchyma with a previously documented intact blood-brain barrier in patients with high grade gliomas.

SECONDARY OBJECTIVE To determine if there is a dose of regadenoson, in the range shown to be safe for clinical administration, that can substantially alter the normalized, contrast enhanced MRI signal intensity in normal-appearing tissues and in: A) Brain adjacent to tumor (i.e. T2 hyperintense, but without contrast enhancement before regadenoson) and B) Contrast enhancing tumor (with contrast enhancement before regadenoson).

Part I Treatment Plan

Part I of the protocol is designed to identify the best regadenoson dose(s) to transiently disrupt the blood-brain barrier as measured by DCE-MRI and contrast enhancement on T1-weighted images corresponding to an increase in the accumulation of MRI contrast (gadolinium) into normal appearing brain contralateral to the brain tumor.

Patients who are at low risk of having complications with a standard regadenoson cardiac stress test (young with no known cardiac disease) and who have had stable MRI scans for at least 2 months prior to enrollment will be asked to undergo a research MRI within two weeks after their most recent previous MRI.

Part II Treatment Plan

Part II will be initiated if the first portion of the study identifies one or more doses of regadenoson that meets the desired endpoint of a Ktrans value >0.04 min-1 within contralateral normal-appearing brain following regadenoson administration. Part II patients will undergo more extensive imaging prior to regadenoson administration to confirm that regadenoson has a significant effect on the BBB using a more comprehensive imaging approach.

Five additional patients who are at low risk to have complications of a standard chemical cardiac stress test (young with no known significant cardiac disease) will be sequentially enrolled at each regadenoson dose meeting the desired endpoint in Part I. In these cohorts, the full research imaging protocol will be utilized in both the pre- and post-regadenoson MRI scans which will allow a direct comparison of all imaging parameters in both the pre-regadenoson and post-regadenoson settings to be directly compared.

ELIGIBILITY:
Inclusion Criteria

1. Patients must have histologically confirmed high grade glioma (including but not limited to glioblastoma (GBM), anaplastic astrocytoma (AA), gliosarcoma, and anaplastic oligodendroglioma). Patients with previous low-grade glioma who progressed after RT/chemotherapy and are biopsied and found to have GBM/GS are eligible.
2. Patients must have measurable contrast-enhancing disease by MRI imaging within 7-14 days of starting treatment (defined by at least 1 cm x 1 cm). Patient must be able to tolerate MRIs with contrast.
3. Patients must have stable MRI (no progression of disease) for the past 2 months or more.
4. Patients may have an unlimited number of prior relapses.
5. The following intervals from previous treatments are required to be eligible:

   * 12 weeks from the completion of radiation.
   * 16 weeks from an anti-VEGF therapy
   * 6 weeks from a nitrosourea chemotherapy
   * 3 weeks from a non-nitrosourea chemotherapy
   * 2 weeks or 5 half-lives from any investigational (not FDA-approved) agents
   * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., erlotinib, hydroxychloroquine, etc.)
6. Age ≥18 years and ≤ 45 years.
7. Karnofsky Performance (KPS) Status 80% (see Appendix A).
8. Patients must have adequate organ and marrow function as defined below:

   - Creatinine ≤ 1.5 mg/Dl or eGFR ≥30 mL/min/1.73 m2
9. Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
10. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of regadenoson are eligible for this trial.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

1. Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
2. Patients who are receiving any other investigational agents.
3. History of hypersensitivity reactions attributed to compounds of similar chemical or biologic composition to regadenoson.
4. Patients with any history, current symptoms, or signs of cardiovascular disease including:

   * any ischemic cardiac event (myocardial infarction, coronary revascularization, stable or unstable angina)
   * Ischemic or nonischemic cardiomyopathy and/or congestive heart failure
   * Supraventricular tachycardia, atrial fibrillation, and/or atrial flutter
   * Ventricular tachyarrhythmias
   * Severe sinus bradycardia defined as a resting heart rate <40 bpm
   * Symptomatic bradycardia, sick sinus syndrome, greater than first-degree AV block, left bundle branch block, and/or presence of a cardiac pacemaker
   * Stenotic valvular heart disease
5. Patients who have uncontrolled hypo- or hypertension defined as a systolic blood pressure <90 mmHg or >180 mmHg, respectively.
6. Patients who have uncontrolled asthma or seizures.
7. Patients taking potential neurotoxic medications - see eligibility criteria of protocol for specific list of medications
8. Patients with uncontrolled concurrent illness.
9. Patients with psychiatric illness/social situations that would limit compliance with study requirements.
10. Pregnant women will be excluded from this study.
11. Because of the potential risk of serious cardiac reactions in the breastfed infant, advise the nursing mother to pump and discard breast milk for 10 hours after administration of regadenoson

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Dose of regadenoson | 15 minutes
  Dose of regadenoson which results in an increase of gadolinium Ktrans by over 10 times.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Grossman, MD, Study Chair — ABTC
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grossman SA, Romo CG, Ye X, Kral B, Strowd RE, Lesser G, Raymond C, Iacoboni M, Desideri S, Fisher J, Danda N, Ellingson BM. Assessing the dose of regadenoson required to transiently alter blood-brain barrier integrity in patients with infiltrating gliomas. Neurooncol Adv. 2025 Feb 15;7(1):vdaf041. doi: 10.1093/noajnl/vdaf041. eCollection 2025 Jan-Dec. PMID 40225909